CLINICAL TRIAL: NCT01893840
Title: Effect on Blood Flow Using the FlowOx™ Device in Patients With Reduced Peripheral Circulation in the Lower Leg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Otivio AS (Industry)
Collaborators: European Union (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OT-FO-01
Record Dates: First submitted 2013-06-26; First posted 2013-07-09 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Periferal Arterial Occlusive Disease, PAOD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FlowOx (Experimental): 5 minutes of pulsating negative pressure (10 sek og -40mmHg/7 sek of athmospheric pressure) will be Applied to the patient's leg
  Interventions: Device: FlowOx

INTERVENTIONS:
Device: FlowOx — Boot-shaped pressure chamber generating pulsating negative pressure

SUMMARY:
A study to assess the effect of negative pulsating pressure therapy on patients with impaired blood flow to the leg caused by arterial disease, to see if the FlowOx device will increase the blood flow to the leg in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Age 30-90 years
* Affected foot/shoe sise less than 46 (approximate foot length less than 29.5 cm)
* Patients with Peripheral Arterial Occlusive Disease (PAOD) grade 2,3 or 4, i.e.:

  1. Clinically verified grade 2, i.e. Intermittent Claudication:

     * Ancle-Brachial Index (ABI)less than 0.9 or
     * Toe brachial Index (TBI) less than 0.7 or
     * Ultrasound and/or CT/Magnetic Resonance (MR) angiography suggesting stenosis(es)and/or occlusion(s)
  2. Clinically verified grade 3, i.e. Critical Limb Ischemia (CLI):

     * ABI less than 0.4 or
     * Toe pressure less than 30 mmHg
     * Rest pain since at least 2 weeks or
     * Use of analgesics for rest pain for at least 2 weeks or
     * Ultrasound and/or CT/Magnetic Resonance (MR) angiography suggesting stenosis(es)and/or occlusion(s)
  3. Clinically verified grade 4, i.e. CLI:

     * Ischemic ulcers or gangrene/tissue loss
     * ABI less than 0.4
     * Toe pressure less than 30 mmHg
     * Rest pain since at least 2 weeks or
     * Use of analgesics for rest pain for at least 2 weeks or
     * Ultrasound and/or CT/MR angiography suggesting stenosis(es)and/or occlusion(s)

Exclusion Criteria:

* Grade 1 PAOD
* Incapable of consenting voluntarily
* Fewer higher than 39 degrees Centigrade
* Severe Chronic Obstructive Pulmonary Disease (COPD)
* Severe heart disease such as unstable angina, severe heart failure and severe valve failure
* Severe Polyneurophathy
* Verified Osteomyelitis other than in the Phanlanx
* Currently treated for cancer and With a life expectancy of less than 2 years

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
% of the prescribed cycles delivered in the specified time FlowOx™-induced change in arterial leg blood flow (LBF) | up to 1 hour
  This is calculated as the difference between the blood flow during the period using FlowOx™ (middle value over a period of 5 minutes) and baseline blood flow (middle value over a period of 5 prior to using FlowOx™)

SECONDARY OUTCOMES:
Patient comfort measured by asking the patient a fixed set of questions | up to 1 hour

OTHER OUTCOMES:
Fitting time | up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Jarlis Wesche, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Akershus University Hospital, Lørenskog, Lørenskog, Norway